CLINICAL TRIAL: NCT05359640
Title: Comparison on Lower Back Pain Treatment: Trigger Bloc vs. Faset Joint Block
Brief Title: Invasive Treatment of Lower Back Pain
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jasmina Markovic Bozic, asist. prof., PhD, University Medical Centre Ljubljana
Other Study IDs: 0120-457/2021/7
Record Dates: First submitted 2022-04-15; First posted 2022-05-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- quality of pain: We will recorded the pain by using a short pain questionnaire and a McGill pain questionnaire.
  Interventions: Other: quality of pain
- consumption of analgesics: The consumption of analgetics, VAS score and improvement of quality of life will be monitored.
  Interventions: Other: quality of pain

INTERVENTIONS:
Other: quality of pain — We will recorded the pain by using a short pain questionnaire and a McGill pain questionnaire.

SUMMARY:
Lower back pain, especially chronic, is a very complex condition that has different causes. There is no single pathophysiological mechanism that could explain the causes of low back pain. It is defined as non-specific and results in only symptomatic treatment. The mechanisms of pain overlap and combine with genetic, epigenetic, individual factors and lifestyle. On the other hand, when low back pain has a defined cause, the treatment can be causal.

At the beginning of the treatment of patients with non-specific low back pain, identification of those that would probably need more complex treatment is tried. More complex patients, are also referred to physiotherapy, and those who are more likely to develop chronic back pain, should be also referred to a psychologist.

An important place, to interrupt the back pain cycle has spine blockades, either local, trigger points blockades, or x-ray-guided blockades of facet joints or nerve roots.

DETAILED DESCRIPTION:
Lower back pain is one of the most common conditions that lead a person to a doctor. It is defined as pain limited upwards by the lower part of the rib arch and down by the lower gluteal crease. It can spread in the lower limb, but not necessarily. About 7.5% of the world's population suffers from back pain. Most people experience an episode of low back pain at least once in their lives. A survey carried out in 2019 on the incidence of chronic pain in Slovenia ranked lower back pain first, with 63% of respondents describing it.

The prevalence of low back pain is between 21% and 75%. In 60% of these individuals it can lead to a reduction in the quality of life due to functional disability. Since 1990, lower back pain has been the leading cause of disability. Causes may be fractures of the osteoporotic vertebrae, spondyloarthritis, malignancy, infections. In 2019, the group of patients aged 50 to 54 were the most affected. Episodes of acute low back pain are usually transient and short-lived, but pain can persists occasionally in more than half of these patients. In most patients with lumbar back pain, the condition improves significantly within six weeks, 33% patients recover within the first three months and in 65% pain remains present also after 12 months. In 33% of patients, the pain recurs within a year after recovery from the previous episode.

Acute and initial chronic (> 6 months) back pain often occurs in the working active population. In 10 percent of patients, acute back pain, lasting more than 6 months, progresses into chronic. After an initial episode, lower back pain often repeates within 12 months after recovery. Treatment should be bio psycho social from the start. The prevalence of back pain is higher in women compared to men (ratio 1.27). This difference is greater when women reach postmenopausal period. It is gender-related (e.g. hormones, differences in the endogenous opioid system). Socio-economic status (level of education) is associated with recurrence of pain and disability, especially in men. The reasons could be behavioural and environmental risks, the professional status, the accessibility to the health system. The socio-economic situation in childhood is a risk factor for the occurrence of back pain in adulthood.

Lower back pain, especially chronic, is a very complex condition that has different causes. There is no single pathophysiological mechanism that could explain the causes of low back pain. Therefore, despite its frequency, we often do not find an exact cause. In 85 - 95% it is defined as non-specific and results in only symptomatic treatment. The mechanisms ob pain overlap and combine with genetic, epigenetic, individual factors and lifestyle. On the other hand, when low back pain have a defined cause, the treatment can be causal. Specific causes of back pain may be fractures, infection, autoimmune diseases, nerve cramping.

Inflammation, hypersensitivity and altered spine innervation are present. Even if nerve tightness due to hernia disci is not present, changes in peripheral nervous system may occur, which may contribute to the development of back pain. The cause could be inflammation in musculoskeletal structures. Compression and degeneration of intervertebral discs are associated with an increase in inflammatory mediators, increased sensory innervation of the disc and plastic changes in peripheral and spinal sensory neuron. These changes indicate a biological mechanism of pain origin. These patients have altered and increased pain sensitivity. This may be due to peripheral or central sensitisation. Hyperalgesia fluctuates with pain intensity and normalises with pain reduction.

According to the latest classification, low back pain is nociceptive, neuropathic or neuroplastic.

In the first case, the pain is caused by irritation of pain-sensing receptors, and in the second by disease or damage of the somatosensory nervous system. In neuroplastic pain perception to stimuli is changed, the patient describes pain, although no clear cause of it is found. When the neuropathic component is also present, pain is more resistant to treatment, the quality of life is even lower and the cost of treatment is higher.

Treatment should be causal when the cause of pain is known. If the neuropathic component is also present then treatment should follow guidelines for neuropathic pain management.

At the beginning of the treatment of patients with non-specific low back pain, identification of those that would probably need more complex treatment was tried. In simple cases education and low doses of simple analgesics are needed. More complex patients are also referred to physiotherapy, and those who are more likely to develop chronic back pain, should be also referred to a psychologist.

An important place to terminate the back pain cycle has spine blockades, either local, trigger points blockades, or x-ray-guided blockades of facet joints or nerve roots.

The research will be conducted in the Department for Chronic Pain, Clinical Department of Anaesthesiology and Intensive Therapy. Patients with chronic low back pain and/or spinal nerve root impairment, scheduled for invasive treatment, will be included in the study. Trigger points blockade were compared to x-ray-guided blockade of small joints of the spine or nerve roots.

Experts from different medical fields are involved in the treatment of chronic low back pain, as the outcome of treatment depends very much on a multidisciplinary approach. Beside the biological component, pain is also affected by the psychological and social components.

In the present research determination after 1, 3 and 6 months after procedure the difference between the groups in pain intensity and in pain quality was tried. The impact of other factors on chronic pain treatment was also determined.

PROTOCOL

In the control group, local anaesthetic and long-acting corticosteroid will be used for trigger blockade. In the study group, a blockade of the small joints of the spine and/or roots of the spinal nerves under x-ray control will also be performed by a combination of local anaesthetic and a long-acting corticosteroid. In each group, 30 patients, will be randomised. The pain will be recorded by using a short pain questionnaire and a McGill pain questionnaire. The consumption of analgesics, VAS score and improvement of quality of life will be monitored.

DATA GHADERING

Following values will be monitored:

* scoring of a Short pain questionnaire and the McGill Pain Questionnaire T
* Analgesic consumption

ELIGIBILITY:
Inclusion Criteria:

* low back pain

Exclusion Criteria:

* under or overage
* pragnancy
* patient refusal

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low back pain, scheduled for invasive approach
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 1 year
  VAS score will be used

SECONDARY OUTCOMES:
improvment of quality of life | 1 year
  McGill pain questionnaire will be used
Pain quality | 1 year
  Short pain questionnaire will be used

CONTACTS AND LOCATIONS:
Overall Officials: Alenka Spindler - Vesel, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] 1. de Souza IMB, Sakaguchi TF, Yuan SLK, et al. Prevalence of low back pain in the elderly population: a systematic review. Clinics (Sao Paulo). 2019;74:e789. Published 2019 Oct 28. doi:10.6061/clinics/2019/e789 2. Makris UE, Abrams RC, Gurland B, Reid MC. Management of persistent pain in the older patient: a clinical review. JAMA. 2014;312(8):825-836. doi:10.1001/jama.2014.9405 3. Hartvigsen J, Hancock MJ, Kongsted A, et al. Series Low back pain 1 What low back pain is and why we need to pay attention. Lancet. 2018;391:2356-2367. doi:10.1016/S0140-6736(18)30480-X 4. Itz CJ, Geurts JW, Van Kleef M, Nelemans P. Clinical course of non-specific low back pain: A systematic review of prospective cohort studies set in primary care. Eur J Pain. 2013;17(1):5-15. doi:10.1002/j.1532-2149.2012.00170.x 5. da C Menezes Costa L, Maher C, Hancock M, McAuley J, Herbert R, Costa L. The prognosis of acute and persistent low-back pain: a meta-analysis. CMAJ. 2012;184(11):1229-1230. doi:10.1503/cmaj.120627 6. Da Silva T, Mills K, Brown BT, Herbert RD, Maher CG, Hancock MJ. Risk of recurrence of low back pain: A systematic review. J Orthop Sports Phys Ther. 2017;47(5):305-313. doi:10.2519/jospt.2017.7415 7. Ferguson SA, Merryweather A, Thiese MS, Hegmann KT, Lu ML, Kapellusch JM, Marras WS. Prevalence of low back pain, seeking medical care, and lost time due to low back pain among manual material handling workers in the United States. BMC Musculoskeletal Disorders. 2019;20:243. 8. Hayden JA, Dunn KM, van der Windt DA, Shaw WS. What is the prognosis of back pain? Best Prac Res Clin Rheumatol. 2010;24:167-179. 9. Da Silva T, Mils K, Brown BT, Pocovi N, de Campos T, Maher C, Hancock MJ. Recurrence of low back pain is common: a prospective inception cohort study. J Physiother. 2019;65(3):159-165. 10. Marin TJ, Van Eerd D, Irvin E, Couban R, Koes BW, Malmivaara A, van Tulder MW, Kamper SJ. Multidisciplinary biopsychosocial rehabilitation for subacute low back pain. Cochrane Database Syst Rev. 2017 Jun 28;6(6):CD002193. 11. Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJEM, Ostelo RWJG, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain: Cochrane systematic review and meta-analysis. BMJ. [7] Dorlin E. L'historicité du sexe. Sexe, genre et sexualités: Presses universitaires de France, 2008. pp. 33-54. 12. Fillingim RB, King CD, Ribeiro-Dasilva MC, Rahim-Williams B, Riley JL, 3rd. Sex, gender, and pain: a review of recent clinical and experimental findings. J Pain 2009;10(5):447-485. 13. Grossschadl F, Stolz E, Mayerl H, Rasky E, Freidl W, Stronegger W. Educational inequality as a predictor of rising back pain prevalence in Austria-sex differences. Eur J Public Health 2016;26(2):248-253. 14. Karran EL, Grant AR, Moseley GL. Low back pain and the social determinants of health: a systematic review and narrative synthesis. Pain 2020;161(11):2476-2493. 15. Lallukka T, Viikari-Juntura E, Raitakari OT, Kahonen M, Lehtimaki T, Viikari J, Solovieva S. Childhood and adult socioeconomic position and social mobility as determinants of low back pain outcomes. Eur J Pain 2014;18(1):128-138. 16. Leresche L. Defining gender disparities in pain management. Clin Orthop Relat Res 2011;469(7):1871-1877. 17. Muthuri SG, Kuh D, Cooper R. Longitudinal profiles of back pain across adulthood and their relationship with childhood factors: evidence from the 1946 British birth cohort. Pain 2018;159(4):764-774. 18. Wang YX, Wang JQ, Kaplar Z. Increased low back pain prevalence in females than in males after menopause age: evidences based on synthetic literature review. Quant Imaging Med Surg 2016;6(2):199-206. 2015;350:h444 19. Wu A, March L, Zheng X, Huang J, Wang X, Zhao J, Blyth FM, Smith E, Buchbinder R, Hoy D. Global low back pain prevalence and years lived with disability from 1990 to 2017: estimates from the Global Burden of Disease Study 2017. Ann Trans Med 2020; 8(6): 299-313. 20. Finucane LM, Downie A, Mercer C, Greenhalgh SM, Boissonnault WG, Pool-Goudzwaard AL, Beneciuk JM, Leech RL, Selfe J. International framework for red flags for potential serious spinal pathologies. J Orth Sports Phys Ther 2020; 50(7): 350-372. 21. Global Health Group Data Exchange http://ghdx.healthdata.org/gbd-results-tool accessed Nov 15, 2020).